CLINICAL TRIAL: NCT05036785
Title: Timing of Suture Removal to Reduce Scarring in Skin Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011060
Record Dates: First submitted 2021-08-26; First posted 2021-09-08 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-09

CONDITIONS: Suture Related Complication

STUDY DESIGN:
Intervention Model Description: Single centre prospective randomized assessor blinded parallel group feasibility study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture removal at 7 days (Active Comparator): Suture removal at 7 days post skin surgery
  Interventions: Other: Timing of suture removal
- Suture removal at 10 days (Active Comparator): Suture removal at 10 days post skin surgery
  Interventions: Other: Timing of suture removal

INTERVENTIONS:
Other: Timing of suture removal — Patients will either be randomized to have their sutures removed at 7 or 10 days post skin surgery

SUMMARY:
This is a single centre prospective randomized assessor blinded parallel group feasibility study that will be undertaken in the Royal Devon and Exeter Dermatology department.

The investigators will be looking at whether timing of percutaneous suture removal after skin surgery impacts on the incidence of suture marks and overall scar cosmesis.

DETAILED DESCRIPTION:
Stitch marks (also known as suture marks or track marks) are permanent marks left in the skin where the stitch has caused local tissue damage and scarring. The risk of these marks is in part thought to be related to the length of time that the stitches are left in place before removal. Stitches are normally left in place for longer on sites where the skin is under greater tension such as the chest or back because there is a concern that the wound may be more likely to open up on these sites. On the chest or back, stitches may be left in place for up to 14 days even though the chest or back is a common site for stitch marks to form.

The investigators are conducting a single centre prospective randomized assessor blinded parallel group feasibility study to estimate a sample size required for a properly powered RCT, and also to provide some preliminary data on the incidence of wound complications and overall scar cosmesis in each group.

All patients attending the dermatology department for wide local excision as part of their skin cancer treatment and primary closure of the subsequent wound will be considered for entry into the trial. Clinicians will identify potential participants during routine practice at their clinic visit. Patients who fulfil the entry criteria will be invited at that appointment to take part.

On the date of participants skin surgery, they will be consented and randomized to either 'suture removal at 7 days' or 'suture removal at 10 days'. Participants will then be booked for a 3 month follow up where the scar site will be evaluated from a patient and clinician perspective to assess suture marks and overall cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years old or above who had capacity to consent to surgery who were willing to attend follow-up appointments within the department

  * Patients undergoing wide local excision as part of their skin cancer treatment pathway
  * Lesions excised from the anterior chest or back
  * Post-operative wound >/= 10mm width
  * Wound could be closed with primary intention healing

Exclusion Criteria:

* Inability to provide valid informed consent and/or unwilling to attend for follow-up

  * Wounds where the edges could not be closely adhered with dermal sutures alone.
  * Wounds requiring a flap or graft for closure.
  * Patients requiring further treatment following original excision eg. Further WLE, radiotherapy etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily McGrath, BMedSci BMBS, Principal Investigator — Royal Devon and Exeter NHS Trust
Locations (1):
- Royal Devon and Exeter Heavitree Hospital, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weitemeyer MB, Bramsen P, Klausen TW, Holmich LR, Gjorup CA. Patient-and observer-reported long-term scar quality of wide local excision scars in melanoma patients. J Plast Surg Hand Surg. 2018 Dec;52(6):319-324. doi: 10.1080/2000656X.2018.1493388. Epub 2018 Oct 31. PMID 30380964
- [Background] Prowse, Phoebe & Shokrollahi, Kayvan. (2014). Leaving our mark - are suture marks acceptable?. Bulletin of The Royal College of Surgeons of England. 96. 264-266. 10.1308/147363514X14042954768637.
- [Background] CRIKELAIR GF. Skin suture marks. Am J Surg. 1958 Nov;96(5):631-9. doi: 10.1016/0002-9610(58)90464-1. No abstract available. PMID 13583327
- [Background] Moy RL, Waldman B, Hein DW. A review of sutures and suturing techniques. J Dermatol Surg Oncol. 1992 Sep;18(9):785-95. doi: 10.1111/j.1524-4725.1992.tb03036.x. PMID 1512311
- [Background] Hasan Z, Gangopadhyay AN, Gupta DK, Srivastava P, Sharma SP. Sutureless skin closure with isoamyl 2-cyanoacrylate in pediatric day-care surgery. Pediatr Surg Int. 2009 Dec;25(12):1123-5. doi: 10.1007/s00383-009-2485-9. Epub 2009 Sep 17. PMID 19760198
- [Background] Hohenleutner U, Egner N, Hohenleutner S, Landthaler M. Intradermal buried vertical mattress suture as sole skin closure: evaluation of 149 cases. Acta Derm Venereol. 2000 Sep-Oct;80(5):344-7. doi: 10.1080/000155500459277. PMID 11200831
- [Background] Wolf R. Serial replacement of sutures for preventing suture marks. J Dermatol Surg Oncol. 1993 Dec;19(12):1131. doi: 10.1111/j.1524-4725.1993.tb02477.x. No abstract available. PMID 8282914
- [Background] Kobayashi S, Ito M, Yamamoto S, Kinugasa Y, Kotake M, Saida Y, Kobatake T, Yamanaka T, Saito N, Moriya Y. Randomized clinical trial of skin closure by subcuticular suture or skin stapling after elective colorectal cancer surgery. Br J Surg. 2015 Apr;102(5):495-500. doi: 10.1002/bjs.9786. Epub 2015 Feb 26. PMID 25727933
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suture Removal at 7 Days | Suture Removal at 10 Days
Started | 30 | 30
Completed | 21 | 18
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture Removal at 7 Days | Suture Removal at 10 Days | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 12 | 7 | 19
Age, Continuous [Mean (Full Range); unit: years] | 66 [24 to 88] | 61 [20 to 88] | 64 [20 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 18 | 39
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Measured Difference in POSAS and VAS Scores Between 7-day and 10-day Groups
Description: In patients undergoing wide local excision and primary wound closure for treatment of skin cancer does earlier removal of percutaneous sutures (7 days rather than 10 days) reduce the incidence of suture marks assessed at 3 months post-operatively.
  The patient and observer scar assessment scale (POSAS) was used. The patient POSAS was comprised of a score between 1-10 each for pain, itch, colour, stiffness, thickness and irregularity.
  The observer POSAS was comprised of a score between 1-10 each for vascularity, pigmentation, thickness, relief, pliability and surface area.
  1 being normal skin and 10 abnormal skin. The total POSAS scores for both patients/observers were calculated by adding these up, with min/max 1-60. Higher scores equating to worse outcomes.
  A visual analogue scale (VAS) was used (min/max 1 to 10) to assess the appearance of suture marks, with 1 being normal skin and 10 being abnormal.
Time Frame: 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Suture Removal at 7 Days | Suture Removal at 10 Days
Number analyzed (Participants) | 21 | 18
score on a scale
  POSAS Total Score (Observer) | 12.9 [6 to 26] | 16.1 [6 to 32]
  POSAS Total Score (Participant) | 19.5 [6 to 44] | 20.3 [6 to 49]
  VAS scores for suture marks (Observer) | 7.2 [3 to 10] | 6.6 [3 to 10]
  VAS scores for suture marks (Participant) | 8.4 [2 to 10] | 7.4 [3 to 10]

2. Secondary Outcome: Does Earlier Suture Removal Have an Impact (Negative or Positive) on Overall Scar Cosmesis and Wound Complication Rates (as Assessed by the Clinician and the Patient)?
Description: The impact on overall scar cosmesis was investigated using the POSAS score (results detailed above) and wound complications rates are detailed below for each group.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Suture Removal at 7 Days | Suture Removal at 10 Days
Number analyzed (Participants) | 21 | 18
participants
  Bleeding | 0 | 0
  Infection | 1 | 2
  Dehiscence | 1 | 1

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events up to 3 months after their procedure.
Description: Patients were given direct contact to the department to voice any concerns over their wound healing. At their 3 month follow up, data was collected to determine whether they had been treated in primary or secondary care for infection/bleeding/dehiscence. This data was self reported by the patient.
Arm/Group | Suture Removal at 7 Days | Suture Removal at 10 Days
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT05036785/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT05036785/ICF_001.pdf